CLINICAL TRIAL: NCT01005797
Title: A Phase I Safety and Tolerability Study of LBH589 in Combination With Sorafenib in Patients With Advanced Renal Cell Carcinoma, Soft Tissue Sarcoma, and Non-small Cell Lung Carcinoma (NSCLC) of Non-squamous Histologies.
Brief Title: Study of Panobinostat in Combination With Sorafenib in Kidney, Soft Tissue or Lung Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101273; CLBH589BUS16T
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Renal Cancer; Non Small Cell Lung Cancer (NSCLC); Soft Tissue Sarcoma
Keywords: Renal Cancer; Non Small Cell Lung Cancer (NSCLC); Solid Tumor; Soft tissue sarcoma; Sorafenib; Panobinostat
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Non-Small-Cell Lung; Sarcoma | interventions — Panobinostat; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Expansion A (Experimental): Expansion A -RCC cohort expansion phase at RP2D: Sorafenib bid daily continuously from cycle 1 (28 day cycle), LBH589 given on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26 of a 28 day cycle.
  Interventions: Drug: Panobinostat (LBH589), Sorafenib
- Expansion B (Experimental): Expansion B -NSCLC cohort expansion phase at RP2D: Sorafenib bid daily continuously from cycle 1 (28 day cycle), LBH589 given on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26 of a 28 day cycle.
  Interventions: Drug: Panobinostat (LBH589), Sorafenib
- Expansion C (Experimental): Expansion C -STS cohort expansion phase at RP2D: Sorafenib bid daily continuously from cycle 1 (28 day cycle), LBH589 on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26 of a 28 day cycle.
  Interventions: Drug: Panobinostat (LBH589), Sorafenib

INTERVENTIONS:
Drug: Panobinostat (LBH589), Sorafenib — Starting dose of sorafenib: 400 mg bid on Day 1-28 of each 28-day cycle; of LBH589: 15 mg on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26 of each 28-day cycle. Administered simultaneously.

SUMMARY:
The purpose of this study is to determine if a new investigational drug called Panobinostat is safe, tolerable and to obtain an initial assessment of efficacy, when given in combination with Sorafenib for the treatment of certain types of lung cancer, kidney cancer and soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old
2. ECOG Performance Status of ≤ 2
3. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
4. Part A (dose escalation): Histologically or cytologically documented metastatic renal cell carcinoma (RCC) of all histologic types, soft tissue sarcoma (STS) limited to the following histologies: angiosarcoma, liposarcoma, and leiomyosarcoma, or non-squamous non-small-cell lung carcinoma (NSCLC). Parts B (RCC) and C (NSCLC) and D (STS)(expanded cohorts). Patients with RCC must have progressive metastatic disease and received at least one multi-kinase inhibitor (e.g., sorafenib/Nexavar or sunitinib/Sutent), or an mTOR inhibitor (e.g., Temsirolimus). Patients with STS must have progressive disease and have received at least two therapeutic regimens (first-line, second-line treatments).

   For patients with metastatic NSCLC, they must have received two standard therapeutic regimens (first-line and second-line treatments).

   In Part A, evaluable disease by radiology and/or a recognized serum tumor marker is required. In Parts B, C, and D measurable disease by RECIST is required
5. Predicted life expectancy ≥ 12 weeks
6. Patients may have had prior therapy, providing the following conditions are met:

   Patients must have recovered from any treatment related toxicities (with the exception of alopecia) to ≤ CTC grade 1 (fatigue, and neurotoxicity at grade 2 are permissible if stable for >3 months) prior to registration.
   1. Chemotherapy: A minimum of 5 predicted half-lives of the agent must have elapsed between the end of treatment and registration on to the study. When halflives are not available the principle of 2 weeks for once daily medications and 3 weeks for agents given less frequently will be adopted, but discussion with the principal investigator is recommended.
   2. Radiation: Patients may have had prior radiation therapy that has not exceeded 25% of bone marrow reserve provided that they have recovered from the acute, toxic effects of radiotherapy prior to registration. A minimum of 7 days must have elapsed between the end of radiotherapy to non-target lesions and registration into the study (minimum of 28 days for target lesions).
   3. Surgery: Previous surgery is permitted provided that wound healing has occurred prior to registration.
7. Patients must meet the following laboratory criteria:

   * Hematology:
   * Neutrophil count of >1500/mm3
   * Platelet count of > 100,000/mm3L
   * Hemoglobin ≥ 9 g/dL
   * Biochemistry:
   * AST/SGOT and ALT/SGPT ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if the transaminase elevation is due to disease involvement
   * Serum bilirubin ≤ 1.5 x ULN
   * Serum creatinine ≤ 2.0 x ULN or 24-hour creatinine clearance ≥ 50 ml/min
   * Total serum calcium (corrected for serum albumin) or ionized calcium ≥ LLN
   * Serum potassium ≥ LLN
   * Serum sodium ≥ LLN
   * Serum albumin ≥ LLN or 2.5 g/dl
   * Patients with any elevated Alkaline Phosphatase due to bone metastasis can be enrolled
8. INR < 1.5 or a PT/PTT within normal limits. Patients receiving anti-coagulation treatment with an agent such as warfarin or heparin may be allowed to participate. For patients on warfarin, the INR should be measured prior to initiation of sorafenib/LBH589 and monitored at least weekly, or as defined by the local standard of care, until the INR is stable. LBH589 and sorafenib may elevate the INR in those on coumadin derivatives
9. Patients must be clinically euthyroid (patients may be on thyroid hormone replacement)'
10. Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal
11. Supportive therapy including bisphosphonates is permissible. Previous use of myeloid and erythroid growth factor support is permissible, but not within 2 weeks of commencement of study. Primary prophylactic use of myeloid and erythroid growth factors is not permitted within the study, but intervention or secondary prophylaxis is permitted if instituted following the documentation of ≥ grade 3 neutropenia or ≥ grade 2 anemia (hemoglobin)
12. Patient must be accessible for repeat dosing and follow-up
13. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of study treatment. and must be willing to use two methods of contraception one of them being a barrier method during the study and for 3 months after last study drug administration

Exclusion criteria:

1. NSCLC of squamous histology.
2. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
3. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
4. Known or suspected allergy to sorafenib or LBH589
5. Impaired cardiac function including any one of the following:

   * Screening ECG with a QTc > 450 msec prior to enrollment to the study
   * Patients with congenital long QT syndrome
   * History of sustained ventricular tachycardia
   * Any history of ventricular fibrillation or torsades de pointes
   * Bradycardia defined as heart rate < 50 beats per minute. Patients with a pacemaker and heart rate ≥ 50 beats per minute are eligible.
   * Patients with a myocardial infarction or unstable angina within 6 months of study entry
   * Congestive heart failure (NY Heart Association class III or IV)
   * Right bundle branch block and left anterior hemiblock (bifasicular block)
6. Uncontrolled hypertension
7. Concomitant use of drugs with a risk of causing torsades de pointes (See Appendix 1.-1)
8. Concomitant use of CYP3A4 inhibitors (See Appendix 1.-2)
9. Patients with unresolved diarrhea > CTCAE grade 1
10. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589
11. Other concurrent severe and/or uncontrolled medical conditions
12. Patients who have undergone major surgery < 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
13. Concomitant use of any anti-cancer therapy or radiation therapy
14. Women who are pregnant or breast feeding or women of childbearing potential (WOCBP)not willing to use a double barrier method of contraception during the study and 3 months after the end of treatment. One of these methods of contraception must be a barrier method. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months).

    Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days of the first administration of oral LBH589
15. Male patients whose sexual partners are WOCBP not using a double method of contraception during the study and 3 months after the end of treatment. One of these methods must be a condom
16. Patients with a history of another primary malignancy within 5 years other than curatively treated CIS of the cervix, or basal or squamous cell carcinoma of the skin
17. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
18. Patients with any significant history of non-compliance to medical regimens or with inability to grant a reliable informed consent
19. Symptomatic brain metastases which are not stable, require steroids, or anti-epileptic medication.
20. Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
21. Pulmonary hemorrhage/bleeding event > CTCAE Grade 2 within 4 weeks of first dose of study drug.
22. Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug.
23. Serious non-healing wound, ulcer, or bone fracture.
24. Use of St. John's Wort or rifampin (rifampicin).
25. Any condition that impairs patient's ability to swallow whole pills.
26. Active or uncontrolled infections, or serious illnesses or medical conditions that could interfere with the patient's ongoing participation in the study.
27. Any other condition, which in the investigator's opinion, would compromise the safety of the patient or the feasibility of completing the study objectives through the use of this patient.

Note: Investigators must ensure that the patients enrolled in the study will be available for all study procedures, including dosing, toxicity assessment and follow up and have the ability to understand the requirements of the study and provide signed informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-11; Primary Completion 2014-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Determine maximum tolerated dose (MTD)for LBH 589 in combination with Sorafenib and establish a recommended phase 2 dose for each drug combination | Point in time when no more than 1 of 6 patients has a Dose Limiting Toxicity (DLT) in cycle 1

SECONDARY OUTCOMES:
Evaluate the safety profile of LGB589 in combination with sorafenib, including DLTs | During the first treatment period (i.e. 28 days) or toxicity similar to DLT after the initial 28-day treatment period
Observe evidence of anti-cancer efficacy estimates of the combination in the tarted expanded cohorts. | Evaluation of disease & re-evaluation for response

CONTACTS AND LOCATIONS:
Overall Officials: Harry Drabkin, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina Hollings Cancer Center, Charleston, South Carolina, United States